CLINICAL TRIAL: NCT00159744
Title: A Phase III, Randomized, Placebo-Controlled, Double-Blind Trial Evaluating the Safety and Efficacy of Sublingual Asenapine vs. Olanzapine and Placebo in In-Patients With an Acute Manic Episode Clinical Trial Protocol 7501004 (Secondary Title: ARES)
Brief Title: 3-Week Study of Asenapine, Olanzapine and Placebo for Treatment of Bipolar Mania (P07008)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P07008; A7501004 (Other: Schering-Plough)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — asenapine; Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Active Comparator): Asenapine
  Interventions: Drug: Asenapine
- Arm 2 (Active Comparator): Olanzapine
  Interventions: Drug: Olanzapine
- Arm 3 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Asenapine — Asenapine, 3 weeks
  Other Names: Org 5222
  Arms: Arm 1
Drug: Olanzapine — Olanzapine, 3 weeks
  Arms: Arm 2
Drug: Placebo — placebo, 3 weeks
  Arms: Arm 3

SUMMARY:
Bipolar disorder is characterized by mood swings that range from high (manic) to low (depressed) states. Sometimes, symptoms of both depression and mania are present (mixed episodes). Asenapine is an investigational medication for the treatment of manic or mixed episodes of bipolar disorder. This is a 3-week study that will test the safety and efficacy of this medication. Patients will receive either asenapine, olanzapine (a medication that is already approved for the treatment of bipolar mania), or placebo (no active medication). Patients will be required to stay in the hospital for at least the first seven days of treatment. Patients that complete the 3 week study may be eligible to continue in extension studies for an additional 9 (study A7501006) to 49 (study A7501007) weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have a DSMIV diagnosis of bipolar I disorder, current episode manic or mixed.

Exclusion Criteria:

* Patients with unstable medical conditions or clinically significant laboratory abnormalities or patients who are rapid cyclers (ie. have had 4 or more (including current) mood episodes in the past 12 months); have any other psychiatric disorder other than bipolar I disorder as a primary diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Actual)
Dates: Start 2004-11-30 (Actual); Primary Completion 2006-04-29 (Actual); Study Completion 2006-04-29 (Actual)

PRIMARY OUTCOMES:
Changes in bipolar manic or mixed symptoms reflected in the scores on the YMRS (Young Mania Rating Scale) | The YMRS was administered at screening, baseline, Day 2, 4, 7, 14 and 21

SECONDARY OUTCOMES:
Ratings on the Clinical Global Impression scale in which severity and improvement of mania, depression, and overall bipolar state are rated. | The CGI assessment at days 1,7 and endpoint (day 21 or the time of the last assessment).
The PANSS (Positive and Negative Symptom Scale) was used to assess psychotic symptoms | The PANSS was administered at Days 1, 7 and 21(or the time of the last assessment).
The MADRS (Montgomery Asberg Depression Rating Scale) was used to assess depressive symptoms | The MADRS was administered on Days 1, 7 and 21(or at the time of the last assessment).l
The Readiness for Discharge Questionaire (RDQ) was administered to characterize the subject's readiness for discharge. The investigator was to make the decision about discharging the subject. | The RDQ was administered on Day 1, 2, 4, 7 , 14 and 21 (or at the time of the last assessment)
CogState, cognition battery, was used to assess changes in cognition | Cog State was administered at screening, Day 1 (baseline) and Days 7, 14, 21 (or endpoint).
SF (short form)-36 and TSQM (Treatment Satisfaction Questionnaire for Medication) -- 2 measures of Quality of Life were administered. | The SF Health Survey was administered at Day 1 and Day 21 or endpoint. The TSMQ was administered at Day 21 or endpoint..
The SARS (Simpson Angus Rating Scale); the AIMS (Involuntary Movement Scale and the BARS (Barnes Akathisia Scale) were used to assess extrapyramidal symptoms | The SARS, AIMS and BARS assessments were administered at Days 1, 7 and 21 or endpoint.
Concomitant medication use was recorded | Concomitant medication use was recorded whenever it occurred
Physical examination, laboratory and electrocardiogram findings and weight/abdominal girth and vital signs were recorded. | Physical exam, ECG, laboratory and weight were recorded at screening and Day 21 or endpoint. Laboratory work was also done at baseline.
Adverse events (AEs) | AEs were recorded whenever they occurred..
Pharmacokinetic analysis was done to determine the level of the drug in the blood | Pk samples were taken at Day 1, 7, 14 and 21 (or endpoint).

REFERENCES:
- [Result] McIntyre RS, Cohen M, Zhao J, Alphs L, Macek TA, Panagides J. Asenapine in the treatment of acute mania in bipolar I disorder: a randomized, double-blind, placebo-controlled trial. J Affect Disord. 2010 Apr;122(1-2):27-38. doi: 10.1016/j.jad.2009.12.028. Epub 2010 Jan 22. PMID 20096936
- [Derived] Suppes T, Eberhard J, Lemming O, Young AH, McIntyre RS. Anxiety, irritability, and agitation as indicators of bipolar mania with depressive symptoms: a post hoc analysis of two clinical trials. Int J Bipolar Disord. 2017 Nov 6;5(1):36. doi: 10.1186/s40345-017-0103-7. PMID 29105003
- [Derived] Michalak EE, Guiraud-Diawara A, Sapin C. Asenapine treatment and health-related quality of life in patients experiencing bipolar I disorder with mixed episodes: post-hoc analyses of pivotal trials. Curr Med Res Opin. 2014 Apr;30(4):711-8. doi: 10.1185/03007995.2013.874988. Epub 2014 Jan 10. PMID 24329543
- [Derived] Szegedi A, Zhao J, McIntyre RS. Early improvement as a predictor of acute treatment outcome in manic or mixed episodes in bipolar-1 disorder: a pooled, post hoc analysis from the asenapine development program. J Affect Disord. 2013 Sep 25;150(3):745-52. doi: 10.1016/j.jad.2013.01.024. Epub 2013 Mar 6. PMID 23473546